CLINICAL TRIAL: NCT04264780
Title: Epilepsy Surgery and Cognition, Psychiatric Function and Quality of Life - Outcome 10 Years or More After Surgery
Brief Title: Epilepsy Surgery and Cognitive Outcome
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Eli Berit Kyte, Psychologist, Oslo University Hospital
Other Study IDs: 651421
Record Dates: First submitted 2019-04-15; First posted 2020-02-11 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: Epilepsy; surgery; temporal lobe
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy | interventions — Neuropsychological Tests; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Younger than 50 years of age: Patients who have undergone epilepsy surgery ten years ago or longer, and are currently less than 50 years of age
  Interventions: Other: Neuropsychological examination
- 50 years of age or older: Patients who have undergone epilepsy surgery ten years ago or longer, and are currently 50 years of age or more
  Interventions: Other: Neuropsychological examination

INTERVENTIONS:
Other: Neuropsychological examination — Neuropsychological follow-up examination, including questionaires
  Other Names: MRI scan

SUMMARY:
This study will give important information about long term consequences of temporal lobe epilepsy surgery on cognition (memory, language, concentration etc), psychiatric function and quality of life.

DETAILED DESCRIPTION:
All patients in Norway who have undergone temporal lobe epilepsy surgery ten years ago or more, will be invited to participate. Two groups will be compared: patients who are younger than 50 years of age vs patients who are older than 50 years of age.

The aim of the study is to improve preoperative information to future epilepsy surgery patients, to aid medical personnel (doctors, psychologists) in the selection of patients for surgery, and to improve knowledge of need for long term follow-up and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Prior temporal lobe epilepsy surgery (10 years ago or more)

Exclusion Criteria:

* Intelligence quotient (IQ) less than 70
* Other main language than Norwegian

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in Norway who have undergone temporal lobe epilepsy surgery ten years ago or more (all of these have also had a preoperative evaluation, including neuropsychological assessment), and who were 20 years of age or older at the time of surgery
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in each study group on neuropsychological tests of memory from baseline (preoperative) to current evaluation | During single data collection session, aproximately 2 hours
  Memory will be measured by Rey Auditory Verbal Learning Test, results reported as raw scores from 1-worst to 15-best; and Diagnosticum für Cerebralschädugung-Revised - DCS-R, results reported as raw scores from 1-worst to 15-best. All results will be converted to T-scores with average 50, standard deviation 10.
Change in each study group on neuropsychological tests of language from baseline (preoperative) to current evaluation | During single data collection session, aproximately 2 hours
  Language will be measured by the subtest "Similarities" from Wechsler Adult Intelligence Scale - WAIS-III, results reported as raw scores from 1-worst to 33-best; Boston Naming Test-results reported as raw scores from 1-worst to 60-best; Letter Fluency from Delis Kaplan Executive Function Scale-D-KEFS, raw scores from 1-worst and up. All results will be converted to T-scores.
Change in each study group on neuropsychological tests of visuospatial abilities from baseline (preoperative) to current evaluation | During single data collection session, aproximately 2 hours
  Visuospatial abilities will be measured by the subtest "Block Design" from WAIS-III, raw scores from 1-worst to 68-best. Results will be converted to T-scores.
Change in each study group on neuropsychological tests of executive function from baseline (preoperative) to current evaluation | During single data collection session, aproximately 2 hours
  Executive function will be measured by the subtest "Digit Span" from WAIS-III, raw scores from 1-worst, to 30-best; Trails A and B from Halstead test battery, raw scores from 1-worst and up. All results will be converted to T-scores.

SECONDARY OUTCOMES:
Score on depression questionaire | During single data collection session, aproximately 2 hours
  Beck Depression Inventory (raw scores divided in 4 categories: 0-13 minimal depression, 14-19 mild depression, 20-28 moderate depression and 29-63 serious depression).
Score on anxiety questionaire | During single data collection session, aproximately 2 hours
  Beck Anxiety Inventory (raw scores divided in 4 categories: 0-7 minimal anxiety, 8-15 mild anxiety, 16-25 moderate anxiety and 26-63 serious anxiety).
Score on quality of life inventory | During single data collection session, aproximately 2 hours
  Quality of Life in Epilepsy - QUOLIE 89 - results will be reported as overall score ranging from 26-worst, to 95-best, and converted to T-score with average 50, standard deviation 10)

CONTACTS AND LOCATIONS:
Overall Officials: Eli B Kyte, Cand.psych, Principal Investigator — OUS - SSE
Locations (1):
- Oslo University Hospital, Spesialsykehuset for epilepsi, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided